CLINICAL TRIAL: NCT00562068
Title: CHOP-Campath, A Pilot Study of CHOP Plus Campath for the Primary Treatment of ALK-ve Peripheral T Cell Lymphoma [CHOP-CAMPATH]
Brief Title: Alemtuzumab and Combination Chemotherapy in Treating Patients With Stage I, Stage II, Stage III, or Stage IV Peripheral T-Cell Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000576439; UCL-BRD/05/170; EU-20785; EUDRACT-2006-000365-11; CTA 21786/0201/001-0001; CRUK-UCL-BRD/05/170-CHOP-CAMPA; UCL-CHOP-CAMPATH
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2008-11

CONDITIONS: Lymphoma; Small Intestine Cancer
Keywords: recurrent adult T-cell leukemia/lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; small intestine lymphoma; peripheral T-cell lymphoma
MeSH Terms: conditions — Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Peripheral | interventions — Alemtuzumab; Cyclophosphamide; Doxorubicin; Prednisolone; Vincristine; Polymerase Chain Reaction; Flow Cytometry

INTERVENTIONS:
Biological: alemtuzumab
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: prednisolone
Drug: vincristine sulfate
Genetic: polymerase chain reaction
Other: flow cytometry
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Monoclonal antibodies, such as alemtuzumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from growing. Giving alemtuzumab together with combination chemotherapy may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of alemtuzumab when given together with combination chemotherapy and to see how well it works in treating patients with stage I , stage II , stage III, or stage IV peripheral T-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the feasibility of adding alemtuzumab to standard cyclophosphamide, doxorubicin hydrochloride, vincristine, and oral prednisolone (CHOP) chemotherapy in patients with stage I-IV peripheral T-cell lymphoma (PTCL).
* To assess the side effect profile and early and late toxicities of this regimen in a standard dose-escalation design, and to establish an appropriate dose level for future studies.

Secondary

* To document response rates and disease-free survival of patients treated with this regimen, and to compare these findings with those of historical controls.
* To monitor immune reconstitution after therapy.
* To determine the pharmacokinetics of subcutaneous alemtuzumab when given in combination with CHOP chemotherapy.
* To more clearly define the CD52 expression profile in these tumors and to investigate phenotypic variations in PTCL.
* To document changes (if any) in levels of Epstein-Barr virus copy number by polymerase chain reaction during CHOP-alemtuzumab therapy.

OUTLINE: This is a multicenter, dose escalation of alemtuzumab study.

Patients receive CHOP chemotherapy comprising cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine IV on day 1 and oral prednisone on days 1-5. Patients also receive alemtuzumab subcutaneously (SC) 1-3 times a week for up to 6 doses per course. Treatment repeats every 3 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo blood collection at baseline, periodically during study treatment, and after completion of study therapy for pharmacokinetics and other correlative studies to monitor cellular immunity. Blood samples are examined by polymerase chain reaction to detect cytomegalovirus antigen and to monitor Epstein-Barr virus copy number. Samples are also analyzed by flow cytometry to quantify circulating B- and T-cells, NK-cells, monocytes, and dendritic-cells.

After completion of study therapy, patients are followed every 3 months for the first year, every 6 months for the second year, and then yearly thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of peripheral T-cell lymphoma (PTCL), including the following subtypes:

  * PTCL not otherwise specified
  * Angioimmunoblastic T-cell lymphoma
  * Anaplastic lymphoma kinase-negative anaplastic large cell lymphoma
  * Intestinal T-cell lymphoma
* Bulky stage IA and stages IB-IV disease (Ann Arbor staging system)
* Expression of CD52 by the tumor
* Measurable or evaluable disease
* No anaplastic lymphoma kinase-positive anaplastic large-cell lymphoma
* No CNS involvement with non-Hodgkin lymphoma

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* No presence of other serious, uncontrolled medical conditions
* No significant anthracycline-related cardiac impairment
* LVEF ≥ 50%
* Creatinine ≤ 1.5 mg/dL
* Bilirubin ≤ 2 times normal value unless due to disease
* Not pregnant or nursing
* Fertile patients must use effective barrier contraception during and for 1 month after completion of study treatment
* No previous malignancy except adequately treated nonmelanoma skin cancer or cervical intraepithelial neoplasia
* No positive serology or non-consenting to test for any of the following:

  * HIV
  * Hepatitis B or C
  * Human T-lymphotropic virus type 1 (HTLV-1)

PRIOR CONCURRENT THERAPY:

* No prior cytotoxic chemotherapy
* Prior radiotherapy may be allowed at the trial coordinator's discretion
* Concurrent consolidation radiotherapy may be given at the clinician's discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Immediate toxicity (incidence of infusion-related reactions)
Hematopoietic toxicity (number of cycles of therapy associated with neutrophils < 0.5e9/L or platelets < 50e9/L)
Incidence of infection (number of days with fever ≥ 38 degrees C, days of intravenous antibiotics, number of inpatient days, number of episodes of cytomegalovirus reactivation)

SECONDARY OUTCOMES:
Disease response (remission rate [complete response and partial response])
Disease outcome (time to progression and overall survival at 2 years from completion of therapy)
Immune reconstitution (time to recover peripheral blood CD4 count to 0.2 e9/L)
Relative dose intensity
Pharmacokinetics assessment of alemtuzumab trough levels before each cycle of treatment
Epstein-Barr virus copy number (measured retrospectively)

CONTACTS AND LOCATIONS:
Overall Officials: Roderick Johnson, MD, Study Chair — Leeds General Infirmary
Locations (5):
- United Kingdom (5):
  - Leeds General Infirmary, Leeds, England
  - King's College Hospital, London, England
  - Royal Marsden - London, London, England
  - Christie Hospital, Manchester, England
  - Torbay Hospital, Torbay Devon, England

REFERENCES:
- [Derived] Phillips EH, Devereux S, Radford J, Mir N, Adedayo T, Clifton-Hadley L, Johnson R. Toxicity and efficacy of alemtuzumab combined with CHOP for aggressive T-cell lymphoma: a phase 1 dose-escalation trial. Leuk Lymphoma. 2019 Sep;60(9):2291-2294. doi: 10.1080/10428194.2019.1576870. Epub 2019 Feb 18. No abstract available. PMID 30773077